CLINICAL TRIAL: NCT04462042
Title: Proton Versus Photon Therapy in Anal Squamous Cell Carcinoma - Swedish Anal Carcinoma Study
Brief Title: Proton Versus Photon Therapy in Anal Squamous Cell Carcinoma
Acronym: SWANCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government); Uppsala County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWANCA
Record Dates: First submitted 2020-06-24; First posted 2020-07-08 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Anal Cancer Squamous Cell
Keywords: proton beam therapy; side effects
MeSH Terms: conditions — Anus Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: The study is an open label, multi-centre, randomised phase II study. 100 patients with anal carcinoma (including carcinoma of the perianal skin) will be randomised in 1:1 ratio to treatment delivered with photons or protons
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photon radiotherapy (Active Comparator): Conventional photon radiation is delivered by volumetric arc therapy/intensity modulated radiotherapy/helical tomotherapy using simultaneous integrated boost (SIB) technique. The total dose to the primary tumour target and node metastases >2 cm is 57.5 Gy in 27 fractions, one fraction/day, five fractions/week during 5.5 weeks. Node metastases up to 2 cm will receive 50.5 Gy in 27 fractions. Elective lymph nodes will receive a total dose of 41.6 Gy.
  Interventions: Radiation: Photon radiotherapy
- Proton radiotherapy (Experimental): Proton radiation is delivered by spot scanning. Proton plans will be produced by single field optimisation/single field uniform dose or multifield optimisation/intensity modulated proton therapy using simultaneous integrated boost (SIB) technique. The total dose to the primary tumour target and node metastases >2 cm is 57.5 Gy(RBE) in 27 fractions, one fraction/day, five fractions/week during 5.5 weeks. Node metastases up to 2 cm will receive 50.5 Gy(RBE) in 27 fractions. Elective lymph nodes will receive a total dose of 41.6 Gy(RBE).
  Interventions: Radiation: Proton radiotherapy

INTERVENTIONS:
Radiation: Proton radiotherapy — Proton radiotherapy
  Other Names: Intensity modulated proton therapy (IMPT)
  Arms: Proton radiotherapy
Radiation: Photon radiotherapy — Conventional photon radiotherapy
  Other Names: Volumetric arc therapy (VMAT), Intensity modulated radiotherapy (IMRT), helical tomotherapy
  Arms: Photon radiotherapy

SUMMARY:
Dosimetric studies suggest that radiotherapy with protons has a potential to reduce side effects compared to treatment with photons for patients with anal carcinoma (AC). There are so far no studies comparing these treatment techniques in a randomised setting. The aim of this study is to compare side effects following photon therapy versus proton therapy within the framework of a randomised controlled trial.

DETAILED DESCRIPTION:
Anal carcinoma is a disease in which modern therapy is reasonably successful in achieving tumour control/cure. Both acute and late side effects are substantial. Proton radiotherapy is hypothesised to have the potential to decrease the incidence/severity of some acute side effects from certain organs at risk e.g. bone marrow and intraperitoneal bowel. By sparing the dose to these organs it is also possible that late effects might be less evident. Sparing of the bone marrow may lead to fewer septic events and dose reductions of chemotherapy which may, as a consequence, improve tumour control. The primary aim of this study is to find ways to decrease acute side effects primarily to alleviate some discomfort from the patient during and after a usually painful treatment experience. It has also been concluded by others that reduction of acute side effects is a relevant aim and end point for the evaluation of new treatment techniques and both patient reported and physician reported data are assessed

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be at least 18 years old
2. Histologically confirmed, previously untreated squamous cell carcinoma (p16-positive or p16-negative) of the anal canal (ICD-O-3 C21), i.e. cancer of the perianal skin without connection to the anal canal are not included. The patients may have primary tumour, regional nodes, metastasis (TNM)-stage T2 (>4 cm) -4,N0-1c,M0 (UICC 8th edition).
3. World Health Organisation/Eastern Cooperative Oncology Group (WHO/ECOG) performance status 0-1
4. The patient must be able to understand the information about the treatment and give a written informed consent.

Exclusion Criteria:

1. Patients with cancer of the perianal skin without involvement of the anal canal (ICD-O-3 C44.5) are not eligible.
2. Patient judged to have any other treatment than radiotherapy with concomitant chemotherapy as the preferred treatment
3. Concomitant or previous malignancies. Exceptions are, adequately treated basal cell carcinoma or squamous cell carcinoma of the skin or, other previous malignancy with a disease-free interval of at least 5 years.
4. Two or more synchronous primary cancers in the pelvic region at time of diagnosis
5. Previous radiotherapy, surgery or chemotherapy that may interfere with the planned treatment for the present disease, as judged by the investigator.
6. Co-existing disease prejudicing survival (expected survival should be >2 years).
7. Pregnancy or breast feeding
8. When prosthetic materials (e.g. hip prostheses) are present close to the target volume it must be considered if this may introduce uncertainties in dose calculations that precludes especially, proton therapy.
9. Patients with pacemaker/ICD are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2031-03-28 (Estimated)

PRIMARY OUTCOMES:
Acute grade >2 hematological side effects | Treatment start until three months after treatment
  Acute hematological side effects will be assessed by weekly full blood cell counts during radiotherapy and the first three weeks after treatment completion. Side Grade >2 acute GI and haematological side-effects during therapy and up to three weeks after the end of treatment. Thereafter, every six weeks for up to three months after treatment. Results will be graded according to the Common Terminology Criteria for Adverse Events (NTCAE) v5.0 scoring system.
  Haematological adverse events will also be assessed by registering febrile episodes during an after treatment as well as the frequency of chemotherapy dose reduction or delayed chemotherapy.

SECONDARY OUTCOMES:
Acute grade >2 gastrointestinal side effects | Treatment start until three months after treatment
  Acute side-effects from the gastrointestinal tract are assess the NTCAE v5.0 scoring system by using. Patient reported side effects are assessed by the European Organization for Research and Treatment of Cancer (EORTC), disease specific quality of life questionnaire for anal cancer, (QLQ-ANL27).
  During radiotherapy, daily reported symptoms will be investigated by a newly developed symptom scale, Radiotherapy related symptom assessment scale (RSAS). The questionnaire includes 13 items specific for current diagnose. The RSAS is a validated instrument for assessing symptom intensity and distress in patients with different cancer disease undergoing radiotherapy, with psychometric properties within the expected range. Answering categories ranges from not at all to a great deal (1-4).
Acute side effects from skin | Treatment start until three months after treatment
  Acute side-effects from skin are assessed by using the Common Terminology Criteria for Adverse Events (NTCAE) v5.0 scoring system. Patient reported side effects are assessed by the European Organization for Research and Treatment of Cancer (EORTC), disease specific questionnaire, QLQ-ANL27.
  During radiotherapy, daily reported symptoms will be investigated by a newly developed symptom scale, Radiotherapy related symptom assessment scale (RSAS). The questionnaire includes 13 items specific for current diagnose. The RSAS is a validated instrument for assessing symptom intensity and distress in patients with different cancer disease undergoing radiotherapy, with psychometric properties within the expected range. Answering categories ranges from not at all to a great deal (1-4).
Acute side effects from the genitourinary tract | Treatment start until three months after treatment
  Acute side-effects from the genitourinary tract are assessed by scoring of genitourinary symptoms, pain by using the Common Terminology Criteria for Adverse Events (NTCAE) v5.0 scoring system. Patient reported side effects are assessed by the European Organization for Research and Treatment of Cancer (EORTC), disease specific questionnaire, QLQ-ANL27.
  During radiotherapy, daily reported symptoms will be investigated by a newly developed symptom scale, Radiotherapy related symptom assessment scale (RSAS). The questionnaire includes 13 items specific for current diagnose. The RSAS is a validated instrument for assessing symptom intensity and distress in patients with different cancer disease undergoing radiotherapy, with psychometric properties within the expected range. Answering categories ranges from not at all to a great deal (1-4).
Pain due to acute radiation reaction | Treatment start until three months after treatment
  Pain is assessed by using the NTCAE v5.0 scoring system. Patient reported pain is assessed by the European Organization for Research and Treatment of Cancer (EORTC), disease specific questionnaire, QLQ-ANL27.
  During radiotherapy, daily reported symptoms will be investigated by a newly developed symptom scale, Radiotherapy related symptom assessment scale (RSAS). The questionnaire includes 13 items specific for current diagnose. The RSAS is a validated instrument for assessing symptom intensity and distress in patients with different cancer disease undergoing radiotherapy, with psychometric properties within the expected range. Answering categories ranges from not at all to a great deal (1-4).
Late side effects from the gastro-intestinal system | From three months after treatment up to five years after treatment
  Late side effects 1, 2 and 5 years after completion of treatment. Side effects from the gastrointestinal system, are assessed by using the NTCAE v5.0 scoring system. Patient reported side effects are assessed by the EORTCs disease specific questionnaire, QLQ-ANL27.
Late side effects | From three months after treatment up to five years after treatment
  Late side effects 1, 2 and 5 years after completion of treatment. Side effects from the genitourinary system are assessed by using the NTCAE v5.0 scoring system. Patient reported side effects are assessed by the EORTCs disease specific questionnaire, QLQ-ANL27.
Late side effects from skin | From three months after treatment up to five years after treatment
  Late side effects 1, 2 and 5 years after completion of treatment. Side effects from the skin are assessed by using the NTCAE v5.0 scoring system. Patient reported side effects are assessed by the EORTCs disease specific questionnaire, QLQ-ANL27.
Assessment of Quality of life (QoL) | From randomisation up to 5 years
  Patient reported quality of life during and after treatment assessed by • HRQoL will be investigated with the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire, the QLQ-C30, supplemented by the disease specific module (anal-cancer) QLQ-ANL27. • EuroQol (EQ-5D) is a generic QoL instrument designed for self-administration. The result could be expressed as a weight with values between zero and one (0-1). Together with information about survival the QoL weight can be expressed as quality-adjusted life-years (QALYs).
Primary tumour response | 3-6 months after treatment
  Frequency of complete tumour regression after primary treatment
Locoregional failure | Up to five years after randomisation
  Time from randomisation until first recurrence, local and/or regional
Disease free survival | Up to five years after randomisation
  Time from randomisation until first recurrence, local/regional/systemic or death
Overall survival | Up to five years after randomisation
  Time from randomisation until death

OTHER OUTCOMES:
Cost-utility analysis | From randomisation until 5 years or death
  Costs and QoL as well as clinical outcome measured as survival time will be considered. The results of the health-economic part of the study will be expressed as cost per quality adjusted life years (QALYs) saved of one intervention in comparison with the other.
  All relevant costs should be identified, quantified, and valued. Also indirect costs related to loss of production when patients cannot work due to the disease.
  All types of resources associated with the two treatment arms during the follow-up should be considered. E.g. costs for treatment of side-effects, costs for surgery when performed, and travelling costs for patients. Costing will be performed at the end of the study.
  For evaluation and analysis of the study results, a relatively simple health-economic model will be developed. This model will be used for evaluation of the two treatment arms from inclusion into the study until 5 years of follow up or death.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Cavalli Björkman, MD, Principal Investigator — Uppsala University Hospital
Locations (4):
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Lund University Hospital, Lund
  - Umeå University Hospital, Umeå
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No
Data may be made available upon request from other researchers to the study group

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT04462042/Prot_SAP_000.pdf